## Stimulant Oxytocin Study

NCT03016598 03/02/2016

## Data Analysis:

Aim 1: We will employ linear mixed effects models to examine within- and betweengroup variability in positive stimulant urine drug screens across 6 weeks.

Aim 2: We will employ linear mixed effects models to examine within- and betweengroup differences in (H2) client and therapist WAI ratings and (H5) attendance rates.

Aim 3: We will use linear mixed effects models to assess within- and between-group differences in the following stress measures related to the Trier Social Stress Test (conducted at baseline and post-6 weeks): (H3) Psychophysiological measures (HR, HRV), (H4) self-reported stimulant craving, (H6) salivary stress biomarkers (cortisol and DHEA), and (H7) self-reported anxiety (STAI-6).